CLINICAL TRIAL: NCT01734148
Title: The RELAX TO SLEEP Study: A Pilot Randomized Controlled Trial
Brief Title: The RELAX TO SLEEP Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Robyn Stremler, Nursing Research Associate, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10000 26217
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Sleep
Keywords: pediatric; sleep difficulties in children; Sleep Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (RELAX TO SLEEP program) (Experimental)
  Interventions: Behavioral: Relax To Sleep Program
- Control group (Usual Care) (No Intervention)

INTERVENTIONS:
Behavioral: Relax To Sleep Program — The educational portion of the program will consist of a standardized educational booklet and a discussion with the PI and provides a brief overview will be given on normal sleep and sleep patterns, children's sleep needs, and the signs and consequences of sleep disturbance. Second, the educational booklet provides sleep hygiene info. The second component consists of of good sleep habits such as having a regular sleep-wake schedule, avoiding caffeine intake prior to sleep, avoiding stimulating activities near nighttime sleep, avoidance of naps during the day, ensuring that the child is exposed to natural light during the day, providing the child with opportunities to socialize during the day. Finally, the program consists of a relaxation breathing technique for the child.
  Arms: Experimental group (RELAX TO SLEEP program)

SUMMARY:
Sleep is a biological process essential for health. Being hospitalized can exacerbate common sleep difficulties in children. Factors that contribute to sleep disturbances during hospitalization include environmental, physiological, and psychological factors. Although sleep interventions exist for healthy children in the community, interventions aimed at hospitalized children need to be developed and piloted with rigorous evaluative methods. The primary purpose of this study is to examine the feasibility and acceptability of the RELAX TO SLEEP program on hospitalized children. Although this study is a pilot study, comparisons will be made to examine sleep outcomes between the intervention group and the control group including: total nocturnal (19h30-07h29), number of nighttime awakenings, longest stretch of nocturnal sleep, and total daytime (07h30-19h29) sleep. Other comparisons include anxiety levels and the development of post-hospital maladaptive behaviours.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 4 and 10.
2. Children expected to stay for 3 nights.
3. Children must have a parent present that plans to stay overnight with the child and must understand English (parent must read English).
4. Child must be in a single private room.

Exclusion Criteria:

1. Children who are receiving palliative care only during their hospital admission.
2. Children diagnosed with a sleep disorder or a clinical anxiety disorder.
3. Children with limited or abnormal movements of both upper and lower extremities (e.g. paralysis, brain injury, cerebral palsy, use of drugs to induce paralysis, musculoskeletal impairments, use of restraints, under heavy sedation), thereby impairing sleep wake activity recording and the inability to use the relaxation breathing exercise.
4. Children who are too acutely ill to participate in the study.
5. Children who have major cognitive impairments that may impact their ability to understand and carry out the intervention.
6. Children who are heavily sedated or receiving benzodiazepines or chloral hydrate.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Total nocturnal sleep at hospital | total measured over 3 days and 3 nights
  Nocturnal sleep in hospital as well as other sleep outcomes will be objectively measured using actigraphy.

SECONDARY OUTCOMES:
Anxiety | Baseline, Day 5
  Anxiety will be measured using the Spence Pre-school anxiety scale for children 4 to 5 years of age , and the Spence Children's Anxiety Scale (SCAS) for children ages 6-10
Post-hospital maladaptive behaviours | Follow-up (5-7 days post discharge)
  member of the research team will make contact within 5-7 days post-discharge by telephone and ask them to complete the Post-Hospital Behaviour Questionnaire (PHBQ), a self-report questionnaire for parents most commonly used for assessing children's post-hospital behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Stremler, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Papaconstantinou EA, Hodnett E, Stremler R. A Behavioral-Educational Intervention to Promote Pediatric Sleep During Hospitalization: A Pilot Randomized Controlled Trial. Behav Sleep Med. 2018 Jul-Aug;16(4):356-370. doi: 10.1080/15402002.2016.1228639. Epub 2016 Sep 15. PMID 27633943